CLINICAL TRIAL: NCT03594175
Title: A Phase 3, Randomized, Double-Blind, Active and Placebo-Controlled Study on the Use of CUSA-081 for Dysfunctional Central Venous Access Devices (CVADs)
Brief Title: Efficacy and Safety of CUSA-081 in the Restoration of Central Venous Access Device (CVAD) Functionality
Acronym: READY1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to ongoing recruitment challenges globally, it is not possible to complete this study. The decision is not based on any reported changes in the safety profile or any concerns with the anticipated efficacy profile of the investigational product.
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUSA-081-HEM-01; 2019-002124-32 (EudraCT Number)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Catheter Occlusion; Thrombosis
Keywords: Central Venous Access Device (CVAD); CUSA-081; reteplase; alteplase; occluded catheters; catheter; occlusion; thrombosis; thrombotic occlusion; CVAD
MeSH Terms: conditions — Thrombosis; Bites and Stings | interventions — reteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CUSA-081 (Experimental): Participants received 1 or 2 doses of CUSA-081, 0.7 milligrams (mg) (0.4 units) per 2 milliliter (mL) directly into the catheter lumen. Participants received the first dose at minute (min) 0, and the second dose (if needed) at min 90.
  Interventions: Drug: CUSA-081
- Placebo (Placebo Comparator): Participants received 1 or 2 doses of placebo (normal saline) directly into the catheter lumen. Participants received the first dose at min 0, and the second dose (if needed) at min 90.
  Interventions: Drug: Placebo
- Alteplase (Active Comparator): Participants received 1 or 2 doses of alteplase, 2 mg/mL, directly into the catheter lumen. Participants received the first dose at min 0, and the second dose (if needed) at min 90.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: CUSA-081 — Participants received 1 or 2 doses of CUSA-081 0.7 mg/2 mL directly into the catheter lumen
  Other Names: Reteplase
  Arms: CUSA-081
Drug: Placebo — Participants received 1 or 2 doses of placebo (normal saline) directly into the catheter lumen
  Arms: Placebo
Drug: Alteplase — Participants received 1 or 2 doses of alteplase, 2 mg/2 mL, directly into the catheter lumen
  Arms: Alteplase

SUMMARY:
To evaluate the efficacy and safety of CUSA-081 (diluted reteplase) in the restoration of central venous access device (CVAD) functionality in participants 18 years and older.

DETAILED DESCRIPTION:
This was a phase III, multinational, multicenter, randomized, double-blind, parallel-group, active and placebo-controlled study to examine CUSA-081 (diluted reteplase) versus placebo or alteplase in subjects with dysfunctional non-hemodialysis Central Venous Access Devices (CVADs).

During the study, the treatment period consisted of 1 visit that may have taken place on the same day as screening or on the following day. After complying with all inclusion criteria, subjects were randomized in a 9:1:6 ratio to CUSA-081 : placebo : alteplase treatment group. A follow-up assessment was performed on Day 30 (±2 days) after treatment with study drug. The end of the study was defined as the last follow-up contact of the last subject to receive study drug in the study.

Routine blood pressure measurement, heart rate and urine pregnancy test were performed before enrolment in the study. Throughout the study, safety assessment included evaluation of treatment emergent adverse events (TEAEs), adverse drug reactions (ADRs), and adverse events (AE) of Special Interest (AESI).

CUSA-081 (reteplase) is a recombinant tissue plasminogen activator (tPA), currently approved in the USA (trade name: RETAVASE®) for treatment of acute ST-elevation myocardial infarction (STEMI) to reduce the risk of death and heart failure.

Alteplase, a biosynthetic form of human tPA, Food and Drug Administration (FDA)-approved under the brand name ACTIVASE® for the treatment of acute ischemic stroke, acute myocardial infarction (AMI) to reduce mortality and incidence of heart failure, and acute massive pulmonary embolism for lysis.

ELIGIBILITY:
Inclusion Criteria:

1. Inability to have 3 mL of blood withdrawn from the selected study catheter;
2. A single or multi-lumen CVAD, implanted ports or peripherally inserted central catheters (PICCs) in place for > 24 hours and documented as previously being patent and functional;
3. Ability to designate one dysfunctional lumen of a multi-lumen catheter to be used throughout the study for both study drug instillation and assessment of CVAD function;
4. Male and non-pregnant female subjects from all racial and ethnic groups 18 years of age and older;
5. Able to have fluids infused at the volume necessary to instil study drug into the CVAD (i.e., up to 2 mL);
6. Informed consent form (ICF) signed and dated indicating that the subject has been informed of and agreed with all pertinent aspects of the study and is willing to comply with all study requirements and procedures.

Exclusion Criteria:

1. CVAD (any type) used for hemodialysis;
2. CVAD known to be dysfunctional for more than 48 hours;
3. Reasonable evidence of mechanical or non-thrombotic occlusion in the selected study catheter (e.g., catheter malposition or migration, sutures, kinks, or precipitates causing obstruction), radiographic assessment is not required;
4. Known or suspected catheter related bloodstream infection (CRBSI);
5. Use of any fibrinolytic agent or anticoagulant (e.g., alteplase, tenecteplase, reteplase, urokinase or heparin) within 24 hours prior to the treatment period (first instillation of study drug). Use of subcutaneous low molecular weight heparin (LMWH) for prophylaxis of thromboembolic events is allowed;
6. Known to be at high risk for bleeding events or embolic complications in the opinion of the Investigator, or has a known condition for which bleeding constitutes a significant hazard (e.g. recent stroke, recent intracranial or intraspinal surgery or serious head trauma, intracranial neoplasm, arteriovenous malformation or aneurysm, known bleeding diathesis);
7. Uncontrolled hypertension (systolic BP ≥160 or diastolic BP ≥110 mmHg) at screening;
8. Clinically unstable in the opinion of the site investigator;
9. Known to be pregnant or breastfeeding at screening;
10. Previously treated in this study (READY 1) or in study READY 2;
11. History of allergic reaction to reteplase, alteplase or vial ingredients (excipients or diluents);
12. Use of any investigational drug or experimental medical device within 28 days prior to treatment; non interventional observational studies participation is allowed.
13. Not mentally, socially, or otherwise able to complete the trial assessment or not likely to survive beyond 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (34):
  - Chiesi Investigational Site, Little Rock, Arkansas
  - Chiesi Investigational Site, Redlands, California
  - Chiesi Investigational Site, Stockton, California
  - Chiesi Investigational Site, Norwich, Connecticut
  - Chiesi Investigational Site, Newark, Delaware
  - Chiesi Investigational Site, Jacksonville, Florida
  - Chiesi Investigational Site, Miami, Florida
  - Chiesi Investigational Site, Plantation, Florida
  - Chiesi Investigational Site, Weeki Wachee, Florida
  - Chiesi Investigational Site, Weston, Florida
  - Chiesi Investigational Site, Atlanta, Georgia
  - Chiesi Investigational Site, Honolulu, Hawaii
  - Chiesi Investigational Site, Quincy, Illinois
  - Chiesi Investigational Site, New Albany, Indiana
  - Einspahr, Topeka, Kansas
  - Chiesi Investigational Site, Lewiston, Maine
  - Chiesi Investigational Site, Hannibal, Missouri
  - Chiesi Investigational Site, Kalispell, Montana
  - Chiesi Investigational Site, Omaha, Nebraska
  - Chiesi Investigational Site, Howell Township, New Jersey
  - Chiesi Investigational Site, New Brunswick, New Jersey
  - Chiesi Investigational Site, Durham, North Carolina
  - Chiesi Investigational Site, Winston-Salem, North Carolina
  - Chiesi Investigational Site, Toledo, Ohio
  - Chiesi Investigational Site, Oklahoma City, Oklahoma
  - Chiesi Investigational Site, Bend, Oregon
  - Chiesi Investigational Site, Portland, Oregon
  - Chiesi Investigational Site, Bethlehem, Pennsylvania
  - Chiesi Investigational Site, Charleston, South Carolina
  - Chiesi Investigational Site, Spartanburg, South Carolina
  - Chiesi Investigational Site, Franklin, Tennessee
  - Chiesi Investigational Site, Knoxville, Tennessee
  - Chiesi Investigational Site, Fredericksburg, Virginia
  - Chiesi Investigational Site, Lynchburg, Virginia
- Argentina (6):
  - Chiesi Investigational Site, Mar del Plata, Buenos Aires
  - Chiesi Investigational Site, Villa María, Córdoba Province
  - Chiesi Investigational Site, Rosario, Santa Fe Province
  - Chiesi Investigational Site, Córdoba
  - Chiesi Investigational Site, Salta
  - Chiesi Investigational Site, San Juan
- Belgium (8):
  - Chiesi Investigational Site, Arlon
  - Chiesi Investigational Site, Bonheiden
  - Chiesi Investigational Site, Bruges
  - Chiesi Investigational Site, Ghent
  - Chiesi Investigational Site, Hasselt
  - Chiesi Investigational Site, Kortrijk
  - Chiesi Investigational Site, Mechelen
  - Chiesi Investigational Site, Roeselare
- Czechia (4):
  - Chiesi Investigational Site, Brno
  - Chiesi Investigational Site, Pilsen
  - Chiesi Investigational Site, Prague
  - Chiesi Investigational Site, Slaný
- Poland (6):
  - Chiesi Investigational Site, Gdansk
  - Chiesi Investigational Site, Katowice
  - Chiesi Investigational Site, Poznan
  - Chiesi Investigational Site, Skawina
  - Chiesi Investigational Site, Tomaszów Mazowiecki
  - Chiesi Investigational Site, Węgrów
- Romania (5):
  - Chiesi Investigational Site, Bucharest
  - Chiesi Invesitgational Site, Cluj-Napoca
  - Chiesi Investigational Site, Constanța
  - Chiesi Investigational Site, Craiova
  - Chiesi Investigational Site, Târgu Mureş
- Spain (3):
  - Chiesi Investigational Site, Terrassa, Barcelona
  - Chiesi Investigational Site, Barcelona
  - Chiesi Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who qualified for the study after completing of all screening assessments were randomized to treatment groups and received the randomized study drug.
Groups:
- CUSA-081: Participants received 1 or 2 doses of CUSA-081, 0.7 milligrams (mg) (0.4 units) per 2 milliliter (mL) directly into the catheter lumen. Participants received the first dose at minute (min) 0, and the second dose, if needed, at min 90.
  CUSA-081: Participants received 1 or 2 doses of CUSA-081 0.7 mg/2 mL directly into the catheter lumen
- Placebo: Participants received 1 or 2 doses of placebo (normal saline) directly into the catheter lumen. Participants will receive the first dose at min 0, and the second dose, if needed, at min 90.
  Placebo: Participants received 1 or 2 doses of placebo (normal saline) directly into the catheter lumen
- Alteplase: Participants received 1 or 2 doses of alteplase, 2 mg/mL, directly into the catheter lumen. Participants received the first dose at min 0, and the second dose, if needed, at min 90.
  Alteplase: Participants received 1 or 2 doses of alteplase, 2 mg/2 mL, directly into the catheter lumen
Period: Overall Study
Arm/Group | CUSA-081 | Placebo | Alteplase
Started | 261 | 28 | 173
Completed | 245 | 25 | 166
Not Completed | 16 | 3 | 7
Not completed — Not treated | 8 | 1 | 5
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline was defined as the last non-missing value available before the first study drug administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | CUSA-081 | Placebo | Alteplase | Total
Number analyzed (Participants) | 253 | 27 | 168 | 448
Age, Categorical [Count of Participants; unit: Participants]
  Age categorical: <=18 years | 0 | 0 | 0 | 0
  Age categorical: Between 18 and 65 years | 140 | 15 | 94 | 249
  Age categorical: >=65 years | 113 | 12 | 74 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.5) | 60.4 (12.7) | 60.9 (14.3) | 60.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 16 | 103 | 269
  Male | 103 | 11 | 65 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: In some countries (e.g. Belgium) it is against the national law to collect information on ethnicity.
  Participants
    number analyzed (Participants) | 177 | 18 | 126 | 321
    Hispanic or Latino | 44 | 7 | 24 | 75
    Not Hispanic or Latino | 132 | 9 | 101 | 242
    Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: In some countries (e.g. Belgium) it is against the national law to collect information on race.
  Participants
    number analyzed (Participants) | 177 | 18 | 126 | 321
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 3 | 1 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 7 | 0 | 5 | 12
    White | 166 | 17 | 119 | 302
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
  kg/m^2 | 28.05 (6.49) | 27.75 (5.62) | 28.01 (6.11) | 28.02 (6.29)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With Treatment Success Following A Single Instillation Of Study Drug With A Dwell Time Up To 90 Min -- CUSA-081 vs Placebo -- Full Analysis Set (FAS)
Description: CUSA-081 vs Placebo -- Single instillation of study drug -- Dwell Time Up To 90 Min -- Full Analysis Set (FAS)
  Treatment success was defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time was up to 90 mins, after a single instillation of study drug. The percentage was calculated as the number of participants with treatment success divided by the total number of participants in the group, multiplied by 100%.
Time Frame: Day 1 (up to 90 mins post dose)
Population: Full analysis set (FAS) was used for the analysis. FAS included all randomized subjects who received at least one dose of study drug, and with at least one available evaluation of efficacy after baseline (i.e., at least one CVAD assessment after study drug administration).
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Placebo
Number analyzed (Participants) | 253 | 27
Participants | 159 | 9
Statistical Analysis 1: Comparison: CUSA-081 vs Placebo; CUSA-081 vs Placebo Dwell Time Up To 90 Min -- FAS; Test type: Superiority; p = 0.003, 2-sample Z test for proportions; Mean difference of proportions, Wald = 29.51, 95% CI 2-sided [10.76 to 48.26]

2. Secondary Outcome: Percentage Of Participants With Treatment Success Following A Single Instillation Of Study Drug With A Dwell Time Up To 90 Min -- CUSA-081 vs Alteplase -- Per Protocol Set (PP)
Description: CUSA-081 vs Alteplase -- Single instillation of study drug -- Dwell Time Up To 90 Min -- Per Protocol set (PP)
  Treatment success was defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time was up to 90 mins, after a single instillation of study drug. The percentage was calculated as the number of participants with treatment success divided by the total number of participants in the group, multiplied by 100%.
  The PP set was used for sensitivity analysis when testing for non-inferiority.
Time Frame: Day 1 (up to 90 min post dose)
Population: Per protocol (PP) set included all subjects from the SAF without any important protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Alteplase
Number analyzed (Participants) | 228 | 152
Participants | 152 | 117
Statistical Analysis 1: Comparison: CUSA-081 vs Alteplase; Test type: Non-Inferiority — Non-inferiority was assessed based on the constructed 95% confidence interval (CI) for the difference in the rate of treatment success between CUSA-081 vs alteplase, with non-inferiority considered as demonstrated if the lower limit of the 95% CI for the difference in rate of success is greater than -10%; p = 0.030, 2-sample Z test for proportions; Mean difference of proportions, Wald = -10.31, 95% CI 2-sided [-19.38 to -1.24]

3. Secondary Outcome: Percentage Of Participants With Treatment Success Following A Single Instillation Of Study Drug With A Dwell Time Up To 60 Min -- CUSA-081 vs Placebo -- Full Analysis Set (FAS)
Description: CUSA-081 vs Placebo -- Single instillation of study drug -- Dwell Time Up To 60 Min -- Full Analysis set (FAS)
  Treatment success was defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time was up to 60 mins, after a single instillation of study drug.
  The percentage was calculated as the number of participants with treatment success divided by the total number of participants in the group, multiplied by 100%.
Time Frame: Day 1 (up to 60 min post dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Placebo
Number analyzed (Participants) | 253 | 27
Participants | 136 | 8
Statistical Analysis 1: Comparison: CUSA-081 vs Placebo; Test type: Superiority; p = 0.017, 2-sample Z test for proportions; Mean difference of proportions, Wald = 24.13, 95% CI 2-sided [5.84 to 42.41]

4. Secondary Outcome: Percentage Of Participants With Treatment Success Following 2 Instillations Of Study Drug With A Dwell Time Up To 180 Min -- CUSA-081 vs Placebo -- Full Analysis Set (FAS)
Description: CUSA-081 vs Placebo -- 2 Instillations of study drug -- Dwell Time Up To 180 Min -- Full Analysis set (FAS)
  Treatment success was defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time was up to 180 mins, following 2 installations of the study drug. The percentage was calculated as the number of participants with treatment success divided by the total number of participants in the group, multiplied by 100%.
  Subjects received the first instillation of study drug (CUSA-081, placebo, or alteplase). If patency was not restored after 90 minutes following the first instillation, a second dose of study drug (the same drug as at first instillation) was administered.
Time Frame: Day 1 (up to 180 min post dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Placebo
Number analyzed (Participants) | 253 | 27
Participants | 207 | 11
Statistical Analysis 1: Comparison: CUSA-081 vs Placebo; Test type: Superiority; p < 0.001, 2-sample Z test for proportions; Mean difference of proportions, Wald = 41.08, 95% CI 2-sided [21.94 to 60.21]

5. Secondary Outcome: Percentage Of Participants With Treatment Success Following A Single Instillation Of Study Drug With A Dwell Time Up To 90 Min -- CUSA-081 vs Alteplase -- Full Analysis Set (FAS)
Description: CUSA-081 vs Alteplase -- Single instillation of study drug -- Dwell Time Up To 90 Min -- Full Analysis set (FAS)
  Treatment success was defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time is up to 90 mins, after a single instillation of study drug. The percentage was calculated as the number of participants with treatment success divided by the total number of participants in the group, multiplied by 100%.
Time Frame: Day 1 (up to 90 min post dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Alteplase
Number analyzed (Participants) | 253 | 168
Participants | 159 | 124
Statistical Analysis 1: Comparison: CUSA-081 vs Alteplase; Test type: Superiority; p = 0.019, 2-sample Z test for proportions; Mean difference of proportions, Wald = -10.96, 95% CI 2-sided [-19.89 to -2.04]

6. Secondary Outcome: Rate Of Recurrent Catheter Dysfunction Within 30 Days Following Treatment With Study Drug
Description: The rate of recurrent catheter dysfunction is defined as re-occlusion. The rate of recurrent catheter dysfunction within 30 days following treatment and the results of the Kaplan-Meier and Cox proportional hazards analyses of the time to first re-occlusion are presented in the FAS.
  This analysis is based on all participants with treatment success following up to 2 administrations of study drug with a total dwell time up to 180 min.
  Subjects received the first instillation of study drug (CUSA-081, placebo, or alteplase). If patency was not restored after 90 minutes following the first instillation, a second dose of study drug (the same drug as at first instillation) was administered.
Time Frame: Day 1 (post dose) up to Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CUSA-081 | Placebo | Alteplase
Number analyzed (Participants) | 207 | 11 | 148
Participants | 17 | 1 | 18
Statistical Analysis 1: Comparison: CUSA-081 vs Placebo; Time to first re-occlusion; Test type: Superiority; Probability Re-Occlusion Free at Day 30 = 0.948, 95% CI 2-sided [0.126 to 7.121]
Statistical Analysis 2: Comparison: CUSA-081 vs Alteplase; Time to first re-occlusion; Test type: Other; Cox Proportional Hazard = 0.654, 95% CI 2-sided [0.337 to 1.270]
Statistical Analysis 3: Comparison: Placebo vs Alteplase; Time to first re-occlusion; Test type: Other; Cox Proportional Hazard = 1.448, 95% CI 2-sided [0.193 to 10.848]

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) Leading to Study Discontinuation
Description: Treatment-emergent AEs leading to study discontinuation were evaluated and the percentage of participants with at least one event reported.
  For all subjects who discontinued the study, the AE was 'Device breakage'.
Time Frame: Day 1 (start of treatment) and until the end of the treatment period (up to 180 min post dose).
Population: The safety set (SAF) included all randomized subjects who received at least one dose of study drug. Subjects discontinued after dosing were included in the SAF.
Measure: Number; unit: % of subjects with at least one event
Arm/Group | CUSA-081 | Placebo | Alteplase
Number analyzed (Participants) | 253 | 27 | 168
% of subjects with at least one event | 1.2 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs) of Special Interest (AESI)
Description: Treatment-emergent AEs of special interest (AESI) were monitored. These included major bleeding (defined as severe blood loss [>5 mL/kg] or blood loss requiring transfusion or causing hypotension requiring use of inotropic agents), embolism, thrombosis, and catheter-related blood stream infection. An adverse event was considered as treatment-emergent if it started on or after the first dose of study drug intake up to the end of the 180-minute treatment period.
Time Frame: Day 1 (start of treatment) and until the end of the treatment period (up to 180 min post dose).
Population: as for outcome 7
Measure: Number; unit: % of subjects with at least one event
Arm/Group | CUSA-081 | Placebo | Alteplase
Number analyzed (Participants) | 253 | 27 | 168
% of subjects with at least one event | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (start of treatment) and until the end of the treatment period (up to 180 min post dose).
Description: Safety set (SAF) was used for the evaluation of AEs.
  SAF included all randomized subjects who received at least one dose of study drug. Subjects discontinued after dosing were included in the SAF.
  Reported are AEs that started on or after the first dose of study drug intake and up to the end of the 180-minute treatment period (treatment-emergent AE).
Arm/Group | CUSA-081 | Placebo | Alteplase
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/27 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/253 | 0/27 | 0/168
Other Adverse Events (participants affected / at risk) | 8/253 | 0/27 | 1/168
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CUSA-081 (N=253) | Placebo (N=27) | Alteplase (N=168)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
13 June 2023, Chiesi issued an initial notification of enrolment hold to all participating study sites for READY 1 study.

05 July 2023, Chiesi issued a voluntary official notification of early termination of study recruitment to all participating sites, due to non-safety reasons. Patient recruitment was slow and completion of the study was not feasible in a reasonable timeframe. Early termination of the study was not expected to impact patient access to other necessary treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03594175/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT03594175/SAP_001.pdf